CLINICAL TRIAL: NCT04592224
Title: Cancer Information Your Way: Get What You Need to Make Your Decisions - a Qualitative Study of Decision Making by Patients With Lower Health Literacy Receiving Care for Incurable Cancer
Brief Title: Cancer Information Your Way: Get What You Need to Make Your Decisions
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 60486
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cancer
Keywords: Health literacy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People diagnosed with cancer may face many difficult decisions regarding their care and preferences. This may be particularly challenging when the cancer cannot be cured. It is therefore hugely important that patients have the information they need so that they can be involved in these decisions and in their care.

This qualitative interview study aims to hear from patients who might have found that the information they were given wasn't easy to understand, or who haven't been able to get involved in their care as much as they would have liked. We hope to learn from these experiences in order to improve the way patients are given information and supported to become involved in their care.

DETAILED DESCRIPTION:
Participants will be identified by healthcare professionals and invited to take part in a single interview either by phone or video call, lasting around an hour.

Interviews will be semi-structured and follow a topic guide, exploring how participants have been given information, how decisions have been made, and any particular challenges they may have faced.

Consent will also be sought for collection of demographic and disease data from the participant's medical record

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of incurable malignancy of any site (as identified by their treating oncologist and may be characterised by eligibility for or receipt of treatment with palliative intent)
* Identified by a member of the healthcare team as potentially having difficulties with health literacy
* Capacity to provide informed consent
* English as the main language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with incurable malignancy of any site, identified by their healthcare professionals as potentially having difficulties with health literacy
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Semi-structured interviews | 1 year
  To explore how best to support decision making by patients with lower health literacy receiving care for incurable cancer, acknowledging the implications COVID-19 will have for future care delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe E Holden, MBBCh, Principal Investigator — Poole Hospital
Locations (1):
- Poole Hospital, Poole, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No